CLINICAL TRIAL: NCT06920446
Title: A Clinical Study Evaluating the Safety and Preliminary Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA in Patients With Relapsed / Refractory Autoimmune Hemolytic Anemia
Brief Title: UCAR T-cell Therapy Targeting CD19/BCMA in Patients With r/r Autoimmune Hemolytic Anemia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Shanghai Xiniao Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-ZY-02
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Relapsed / Refractory Autoimmune Hemolytic Anemia
Keywords: Universal Allogeneic CAR T-cells; CD19/BCMA CAR T-cells
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-CD19/BCMA CAR T-cells (Experimental): UCAR T-cell group
  Interventions: Biological: UCAR T-cell group

INTERVENTIONS:
Biological: UCAR T-cell group — A single injection of UCAR T-cells, referred to as universal allogeneic anti-CD19/BCMA CAR T-cells

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with relapsed or refractory Autoimmune hemolytic anemia. This study aims to evaluate the safety and efficacy of the treatment with universal CD19/BCMA CAR T-cells.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal CD19/BCMA CAR T-cells in Relapsed or Refractory Autoimmune hemolytic anemia.

Study intervention consists of a single infusion of universal CAR T-cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

Interim analysis will be performed when participants finish the visit 90 days after CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Flow cytometry detected positive B cell CD19 or BCMA in the patient's peripheral blood.
3. Patients diagnosed with AIHA, including warm antibody type, cold agglutinin disease, mixed type, and other types of AIHA, with diagnostic criteria referring to the "Chinese Adult Autoimmune Hemolytic Anemia Diagnosis and Treatment Guidelines (2023 Edition) .
4. The definition of recurrent/refractory AIHA that has received at least 3 failed lines of treatment is symptomatic anemia (hemoglobin<100g/L) that persists after a routine treatment cycle of at least 6 months and is still ineffective or reappears after disease remission. The definition of conventional treatment: treatment with glucocorticoids and/or rituximab, as well as any 1-2 or more of the following immunomodulatory drugs: cyclophosphamide, azathioprine, mycophenolate mofetil, cyclosporine A, azathioprine, danazol, bendamustine, fludarabine, bortezomib, and biologics including daratumumab, BTK inhibitors, Syk inhibitors, and complement inhibitors.
5. Functional requirements for major organs are as follows:

   1. The bone marrow function needs to meet: a Neutrophil count ≥ 0.5× 10 ^ 9/L; b. Platelets ≥ 30 × 10 ^ 9/L.
   2. Liver function: ALT ≤ 3 × UL; AST ≤ 3×ULN.
   3. Renal function: creatinine clearance rate (CrCl) ≥ 30 ml/min (Cockcroft/Gault formula).
6. ECOG ≤ 2
7. Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative Human chorionic gonadotropin (HCG) test within 7 days before study enrollment and not be lactating.
8. Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Subjects with a history of severe drug allergies or allergic tendencies.
2. Presence or suspicion of uncontrolled or treatment-required fungal, bacterial, viral, or other infections.
3. Subjects with central nervous system diseases caused by autoimmune diseases or non-autoimmune diseases (including epilepsy, psychosis, organic brain syndrome, cerebral vascular accidents, encephalitis, central nervous system vasculitis).
4. Subjects with insufficient cardiac function.
5. Subjects with congenital immunoglobulin deficiencies.
6. History of malignancy within five years.
7. Subjects with end-stage renal failure.
8. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titer higher than the upper limit of detection; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV) antibody; individuals positive for syphilis testing.
9. Subjects with psychiatric disorders and severe cognitive impairments.
10. Subjects who have used immunosuppressive agents or biologics with therapeutic effects on the disease within five half-life before enrollment.
11. Pregnant women or women planning to conceive.
12. Active infection, active rheumatic and immune disease, drug induced and diagnosed lymphoproliferative tumor associated secondary AIHA patients.
13. Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The number and severity of dose-limiting toxicity (DLT) events | Within 28 Days After UCAR T-cell Infusion
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells.
The total number, incidence, and severity of AEs | Up to 90 days After UCAR T-cell Infusion
Clinical response | Up to 24 Months After UCAR T-cell Infusion
  Rates of CR, CRi, PR, ORR